CLINICAL TRIAL: NCT00961376
Title: Vaccination of Chemotherapy Induced Lymphopenic Unresectable Stage III or Stage IV Melanoma Patients Following Reconstitution With Total or CD25-depleted PBMC
Brief Title: Vaccination of Melanoma Patients With Total or CD25-depleted Peripheral Blood Mononuclear Cell (PBMC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Discretion
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHS IRB 06-55
Record Dates: First submitted 2009-08-14; First posted 2009-08-19 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Melanoma
Keywords: melanoma; unresectable stage III or IV melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Active Comparator): PBMC re-infusion
  Interventions: Biological: PBMC re-infusion
- Cohort B (Experimental): CD25 depletion
  Interventions: Biological: CD25 depletion

INTERVENTIONS:
Biological: PBMC re-infusion — Autologous PBMC re-infusion
  Arms: Cohort A
Biological: CD25 depletion — Autologous, CD25-depleted PBMC re-infusion
  Arms: Cohort B

SUMMARY:
The objective of this study is to evaluate the safety and immunologic effects of autologous tumor vaccination administered with human granulocyte-macrophage colony-simulating factor (hGM-CSF), and subsequent boosting vaccinations in patients made lymphopenic by treatment with chemotherapy and infused with autologous PBMC (Cohort A) or CD25 depleted PBMC (Cohort B). Clinical observations and laboratory measurements will be monitored to evaluate safety, toxicity, immune responses, and anti-tumor effects. Additionally, the effects of treatment on tumor response will be evaluated.

DETAILED DESCRIPTION:
This is an open-label, outpatient Phase II, prospective, randomized, single-center, clinical trial. Up to 14 patients with a diagnosis of unresectable stage III or stage IV melanoma.

All patients will undergo leukapheresis to collect PBMC.

All patients will receive Cyclophosphamide 350 mg/m2 dl-3 and Fludarabine 20 mg/m2 dl-3.

Following chemotherapy to induce lymphopenia, patients will be re-infused with PDMC as follows:

Autologous PBMC re-infusion (Cohort A) Autologous, CD25-depleted PBMC re-infusion (Cohort B)

Following PBMC re-infusion, all patients will receive subcutaneous GM-CSF Infusion (50 micrograms/24 hrs) continuously for 6 days.

All patients will then receive 4 booster vaccinations as follows:

Intradermal injection of autologous tumor cells in the lower abdomen to deliver a total dose of at least 2x107 cells administered week 3, week 5, week 9 and week 13. Subcutaneous GM-CSF Infusion (50 micrograms/24 hrs) adjacent to the vaccine site begins at time of vaccination (week 3, 5, 9 and 13) and continues for 6 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed malignant melanoma that is unresectable stage III or stage IV. Measurable disease is not required.
* Patients must have failed, refused, or not been eligible to receive at least one standard therapy regimen for metastatic disease.
* Easily harvested metastatic tumor cells e.g., skin or lymph node metastases or a planned surgery to remove tumor. Patients undergoing resection of a solitary brain metastasis are eligible if their resected lesion contains an adequate number of tumor cells. A minimum 2 cm x 2 cm x 2 cm lesion will be required for study eligibility.
* Sufficient viable tumor cells harvested to generate the vaccine. The tumor collected must contain greater than 1.6 x 108 viable tumor cells or a cell line generated from autologous tumor must provide greater than 1.6 x 108 viable tumor cells.
* Patients may have received prior chemotherapy and/or immunotherapy. Prior radiation therapy is acceptable but previously radiated sites may not be used for tumor collection for vaccine preparation.
* Life expectancy of greater than or = 3 months.
* ECOG performance status <2 (Karnofsky >60%; see Appendix A).
* Patients must have normal organ and marrow function at the time of enrollment as defined in the protocol.
* Patients must be seronegative for HIV, Hepatitis B surface antigen and Hepatitis C antibody.
* If patients have had recent surgery, they must have recovered from the effects of that surgery in the opinion of the investigator.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C).
* Radiation therapy within 2 weeks. Prior radiation must have been to less 30% of the bone marrow and patient has recovered from all side effects, in the opinion of the investigator.
* Patients may not be receiving any other investigational agents.
* Steroid therapy, other than replacement steroids and inhaled steroids. Patients who might require systemic corticosteroids other than replacement steroids during the next three months are not eligible for this study.
* Patients with known brain metastases unless treated with radiation therapy and/or surgery and shown to be stable > 1 month.
* Autoimmune disease requiring treatment, with the exception of controlled autoimmune thyroiditis or vitiligo.
* Pregnant or nursing women are excluded from this study because fludarabine and cyclophosphamide have potential teratogenic effects. It is not known whether fludarabine is excreted in breast milk but the package insert cautions that it might and recommends against breastfeeding if the mother is treated with fludarabine.
* Uncontrolled intercurrent illness which, in the opinion of the investigator, may increase the risks associated with study participation or interfere with the interpretation of the results..
* Any other medical illness or psychiatric condition/social situations that in the opinion of the principal investigator would compromise the patients ability to tolerate this treatment or would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-02-10 (Actual)

PRIMARY OUTCOMES:
Immunologic effects (changes in the number of tumor specific T cells) | Up to day 119
  The absolute number and frequency of tumor specific T cells will be measured at days 7, 21, 35, 64, 91, and day 119.

SECONDARY OUTCOMES:
The number and severity of adverse events | Up to day 119
  Adverse events will be assessed on Days 7, 21, 35, 64, 91, and 119. Of special interest will be any adverse events thought to represent an autoimmune reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Curti, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States